CLINICAL TRIAL: NCT05062915
Title: Diagnostic Work up and Management of Acute Onset Vertigo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Helle Elisabeth Agger-Nielsen, Doctor, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20/12302
Record Dates: First submitted 2021-09-08; First posted 2021-09-30 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Acute Vestibular Syndrome; Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Intervention Model Description: Step 1:A prospective cohort of patients with acute Vestibular Syndrome (AVS) is compared to a baseline (historical) cohort. For a period of 1 year all patients with AVS are registred (baseline population 1) after 1 year their chart is reviewed and those with peripheral AVS (baseline population 2) are invited for a follow up. Those patients in the baseline population 2 who still has a balancedeficit are offered late onset vestibular rehabilitation.
  Step 2: all patients admitted with AVS are enrolled as Study population 1, all have balancetesting (V-HIT, HINTS, Posturography and MRI) done upfront. From study population 1, the patients with peripheral AVS (study population 2) are offered (besides the workup with V-Hit and MRI) a vestibular rehabilitation programme (early onset rehabilitation).
Masking Description: Bloc randomisation done by a physical therapist: only for the part of the study with vestibular rehabilitation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline population (No Intervention): Historic cohorte for comparisson in study 1. Baseline population 1 all patients with AVS. Baseline 2 population part of baseline 1 but with peripheral cause of AVS. Are offered late onset vestibular rehabilitaion if they have balance deficit.
- Study population (Active Comparator): The study population is divided into 2 groups, based on the findings in the clinical investigation.
  study population 1: all patients with acute Vestibular syndrome (AVS) Study population 2: all patients from study group 1, with vestibular/peripheral cause of AVS. They are offered early onset rehabilitation.
  Arm 1 and 2 are compared for cost-effectiveness and compared to the costs of the diagnosis.
  Interventions: Diagnostic Test: HINTS

INTERVENTIONS:
Diagnostic Test: HINTS — HINTS (Head Impulse, Nystagmus, test of skew) V-HIT (Head impulse test google assisted) MRI: 3-4 MRI of the brain including the posterior fossa Vestibular rehabilitation for all patients with a vestibular deficit.
  Other Names: V-VHIT; MRI
  Arms: Study population

SUMMARY:
Incidence: Dizziness or vertigo is a very prevalent complaint in the general population, and a common reason for seeking medical attention. In Denmark, 20-30 % have experienced dizziness/vertigo to a degree that has led to disability, sick leave, or medical contact(1). In the United States, dizziness is estimated to account for partly 2.6-4.4 million visits to emergency departments (EDs) each year, partly 4 % of main symptoms in patients admitted to EDs (2). In Germany, the estimated prevalence of dizziness is 20-30 % with an annual incidence about 11 % (3).

Terminology and definition: Dizziness or vertigo is not a disease itself but rather a symptom of various underlying disorders. Thus, vestibular, neurological, cardiovascular, metabolic, and psychiatric diseases may be associated with dizziness/vertigo as well as medical side effects. Patients (and professionals) often use the two terms dizziness and vertigo synonymously, which may cause some confusion in the choice of diagnostics. Vertigo is characteristic for vestibular disorders and is defined as sensation of self-motion when no self-motion occurs, or sensation of distorted self-motion during an otherwise normal head movement, whereas dizziness is a feeling of more general unsteadiness.

1. Is implementation of HINTS and v-HIT in an ED able to reduce the number of undiagnosed and misdiagnosed cases of acute onset vertigo as well as diagnostic delay ?
2. What are the effects of immediate and systematic balance training in case of acute vestibular diseases ?
3. What is the cost-effectiveness of implementation of HINTS and v-HIT as up front diagnostics, and systematic balance training in patients with acute vestibular diseases ?

DETAILED DESCRIPTION:
Phd thesis will be done including these 3 parts. STUDY 1 Effects of implementation of HINTS and v-HIT in an emergency department HYPOTHESIS Implementation of HINTS and v-HIT in the acute diagnostic workup for patients presenting with acute onset dizziness/vertigo at the ED, Hospital of South West Jutland (SVS), Denmark, along with the routine triage and acute MRI of the brain can reduce the number of un-/misdiagnosed cases to almost zero at the time of discharge from hospital.

HINTS and V-hit can be performed by a nurse at the ED with a high level of accuracy.

AIMS To investigate the effects of implementing nurse-performed v-HIT and HINTS in patients presenting with acute onset dizziness/vertigo in the ED.

DESIGN A prospective cohort of unselected patients with acute onset dizziness/vertigo is compared to a baseline (historical) cohort.

POPULATIONS

Two populations are included:

Baseline population 1 (historical cohort being identified by reviewing charts of all consecutive patients in the ED throughout 12 months prior to implementation of intervention 1.

Study population 1: all consecutive patients undergoing intervention 1 (prospective cohort) throughout 12 months. Inclusion criteria: all consecutive adult patients (18 years and older) admitted to the ED with acute onset vertigo/dizziness as the primary complaint. Exclusion criteria: patients with known vestibular disease, vestibular symptoms lasting more than two days.

Two hundred patients are needed in both groups (see sample size calculation in the statistical section).

METHODS Baseline population 1: The first part of this study reviews the patient's pathway from onset of vertigo/dizziness to final diagnosis by means of current management. Charts of all patients admitted to the ED, SVS, throughout 12 months due to acute onset dizziness/vertigo as the primary complaint are reviewed. Data is used for comparison with study population 1 undergoing intervention 1. In addition, the baseline population are offered a cross sectional follow up visit at the ENT Department, SVS, in order to fill in DHI (Dizziness Handicap Inventory), as well as undergoing standard vestibular status with HINTS, v-HIT, VNG (spontaneous nystagmus) and posturography. A subgroup of baseline patients with assumed peripheral AVS at the time of the acute attack is appointed according to patient chart, actual history and vestibular status as baseline in study 2 (baseline population 2).

Study population 1: is enrolled prospectively and represents all consecutive patients admitted with acute onset dizziness/vertigo as the primary complaint to the ED. The population undergoes intervention 1: HINTS and v-HIT performed acutely by a group of trained nurses in the ED. Furthermore, acute MRI and usual triage is performed.

Intervention 1: The group of 5-6 nurses at the ED is trained by two experienced ENT specialists performing HINTS, v-HIT, and VNG (spontaneous nystagmus). After a month of five training sessions, the nurses perform the examinations at the ED. All tests results including MRI and routine triage are conferred with the senior doctor on duty in the ED, and it is decided to which specialty the patient is referred. HINTS, v-HIT, and VNG are repeated at the ENT Department within 24 hours to investigate the accuracy of the primary findings in the ED. Patients with peripheral AVS are identified in order to be included in study 2 with intervention 2 (study population 2).

Comparability of the baseline population and study population 1 will be performed by demographics.

PRIMARY OUTCOMES Number of undiagnosed and misdiagnosed cases in the two populations is calculated at the time of discharge from ED. Definitions: Undiagnosed: cases without specific ICD10 code explaining acute dizziness/vertigo. Misdiagnosed: cases in which the chart review (baseline population) reveals obviously wrong ICD10 codes/post-hospital examinations reveal the specific cause of dizziness/vertigo; or ENT-examination within 24 hours changes the primary diagnosis (study population 1).

Percentage of patients undergoing HINTS in the baseline population, and percentage of patients undergoing HINTS and v-HIT in study population 1.

SECONDARY OUTCOMES Time to correct diagnosis. Primary referral to relevant specialty: internal medicine, cardiology, neurology, or ENT: number of correct referrals from ED. Accuracy of nurse-performed HINTS and v-HIT using the results of ENT specialist-performed HINTS and v-HIT as reference.

VARIABLES Age, gender, level of education, work, nutritional-, smoking-, alcohol-, and exercise factors (equivalent of the Danish KRAM factors), BMI, examinations and number hereof, comorbidities, previous vertigo/dizziness, medication, time to ICD diagnosis after admittance (hours), diagnosis, correctness of diagnosis evaluated at follow up at the ENT Department (right/wrong/no initial diagnosis)., HINTS (normal, not normal, not done), v-HIT (video head impulse (lateral): gain after 60 ms, gain asymmetry (%), saccades overt and covert), VNG (spontaneous nystagmus, fixed and unfixed gaze).

Based on the ENT examination a subgroup of study population 1 suffering from peripheral AVS is enrolled in study 2 undergoing intervention 2: rehabilitation.

STUDY 2 Effects of immediate and systematic balance training in patients with peripheral acute vestibular diseases.

HYPOTHESIS Patients suffering from any peripheral AVS: vestibular neuritis, benign paroxysmal positioning vertigo (BPPV), debut of Meniere's disease, perilymphatic fistulas, vestibular migraine, or labyrinthitis benefit from targeted vestibular balance training.

AIM The objective is to investigate the number of patients regaining complete balance after peripheral AVS and to compare a historical group undergoing no balance training with a prospective cohort undergoing systematic balance training immediately after the acute attack.

DESIGN Prospective, comparative interventional study. POPULATIONS Baseline population 2: patients identified as baseline population 1 will be contacted 12 months after the acute admission to ED for a vestibular status at the ENT Department. Those suspected of having suffered from any kind of peripheral AVS at the time of the acute attack according to the chart, actual history and vestibular status will be invited to go through the same balance training and follow up as study population 2.

Study population 2 is generated based on the findings in study population 1: those diagnosed with peripheral AVS according to the ENT examinations (vestibular status within 24 hours after admission) are offered a systematic and structured balance training program.

One hundred patients are needed in both groups (see sample size calculation in the statistical section).

Comparability of the two populations will be examined by demographics. METHODS Vestibular status: DHI, HINTS, v-HIT, VNG, and posturography. Intervention 2: The balance training program consists of a six step gaze stabilizing exercise program and a four step general balance stabilizing exercise program, introduced as soon as the patient is able to stand on their own. The progress of the program is evaluated by DHI and posturography in the outlined time intervals. The programs are individualized so each step is mastered before moving on to the next step. Patients will be instructed by a physiotherapist and/or a trained nurse in continuation of going through the vestibular status at the ENT Department.

Follow up: Progress with the program is evaluated with vestibular status once a week for six weeks and then after, three, six and twelve months for a final evaluation.

PRIMARY OUTCOMES Percentage of patients with complete recovery one year after the acute attack defined as resumption of all daily day activities. Degree of vestibular deficit scored by the DHI questionnaire. Vestibular status in baseline population 2 (12 months after admission) is compared to vestibular status at one year follow up in study population 2 in terms of HINTS, v-HIT, VNG, posturography.

SECONDARY OUTCOMES Vestibular status in study population 2 at admission and at one year follow up are compared. Progression through the balance training program is evaluated by change in vestibular status.

VARIABLES Age, gender, level of education, work, nutritional-, smoking-, alcohol-, and exercise factors (equivalent of the Danish KRAM factors), BMI, comorbidity, previous vertigo/dizziness, medication, history of substance abuse. DHI (points), HINTS (normal, abnormal), v-HIT (video head impulse (lateral): gain after 60 ms, gain asymmetry (%), saccades overt and covert), VNG (spontaneous nystagmus, fixed and unfixed gaze), posturography (degrees of sway measured in different positions: standing, standing closed eyes, standing on pillows).

STUDY 3 Cost-effectiveness of implementing up front diagnostics and balance training in patients with acute onset dizziness.

HYPOTHESIS Changes of up front diagnostics in patients with acute onset dizziness/vertigo as well as implementation of balance training is associated with increased costs. However, such improvements result in higher percentage of patients with complete recovery and an earlier return to work and thereby reduces the total socio-economic burden related to the incident.

AIM To examine the cost-effectiveness of up front diagnostics and balance training in prospective cohorts of patients with acute onset dizziness compared to a historical control group.

POPULATIONS Baseline population 1, study population 1, baseline population 2 and study population 2.

METHODS A cost-effectiveness analysis will be conducted from a societal perspective with one year follow-up. Total costs of all patients will be measured, valued, and analysed. In the analysis, the difference in cost will be related to percentage of patients with complete recovery one year after the acute attack.

Costing: The costs of up front diagnosis and balance training will be estimated using micro-costing. Use of primary healthcare services (including costs to general practitioner, specialized doctor, physiotherapist, etc.) will be extracted and valued from the Danish National Health Service Register for Primary Care (NHSR). Use of secondary healthcare services will be extracted from the National Patient Registry (NPR). This register includes information on hospital departments, dates of admission and discharge, and diagnosis. The valuation is determined by reimbursement rates from the Diagnosis-Related-Grouping (DRG) and the Outpatient-grouping-system (DAGS). Productivity loss will be extracted from the Danish Register for Evaluation of Marginalization (DREAM) and valued by age- and gender-matched average gross salaries from Statistics Denmark (www.dst.dk).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: all consecutive adult patients (18 years and older) admitted to the ED with acute onset vertigo/dizziness (AVS) as the primary complaint.

Exclusion Criteria:

* patients with known vestibular disease, vestibular symptoms lasting more than two days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of undiagnosed and misdiagnosed cases | 1,5 years
  cases in the two populations is calculated at the time of discharge from ED. Definitions: Undiagnosed: cases without specific ICD10 code explaining acute dizziness/vertigo. Misdiagnosed: cases in which the chart review (baseline population) reveals obviously wrong ICD10 codes/post-hospital examinations reveal the specific cause of dizziness/vertigo; or ENT-examination within 24 hours changes the primary diagnosis (study population 1).
Percentage of patients undergoing HINTS in the baseline population | 1 year
  Percentage of patients undergoing HINTS in the baseline population, and percentage of patients undergoing HINTS and v-HIT in study population 1.
Percentage of patients with complete recovery | 1,5 years
  Percentage of patients with complete recovery one year after the acute attack defined as resumption of all daily day activities. Degree of vestibular deficit scored by the DHI questionnaire. Vestibular status in baseline population 2 (12 months after admission) is compared to vestibular status at one year follow up in study population 2 in terms of HINTS, v-HIT, VNG, posturography.
Cost-effectiveness of implementing up front diagnostics and balance training in patients with acute onset dizziness | 1 years
  To examine the cost-effectiveness of up front diagnostics and balance training in prospective cohorts of patients with acute onset dizziness compared to a historical control group. A cost-effectiveness analysis will be conducted.
  Costing: The costs of up front diagnosis and balance training will be estimated using micro-costing. Use of primary healthcare services will be extracted and valued from the Danish National Health Service Register for Primary Care (NHSR). Use of secondary healthcare services will be extracted from the National Patient Registry (NPR). Productivity loss will be extracted from the Danish Register for Evaluation of Marginalization (DREAM) and valued by age- and gender-matched average gross salaries from Statistics Denmark (www.dst.dk).

SECONDARY OUTCOMES:
Time to correct diagnosis | 1,5 years
  Time to correct diagnosis. Primary referral to relevant specialty: internal medicine, cardiology, neurology, or ENT: number of correct referrals from ED. Accuracy of nurse-performed HINTS and v-HIT using the results of ENT specialist-performed HINTS and v-HIT as reference.
Vestibular status in study population 2 at admission and at one year follow up are compared. Progression through the balance training program is evaluated by change in vestibular status | 2,5 years
  Vestibular status in study population 2 at admission and at one year follow up are compared. Progression through the balance training program is evaluated by change in vestibular status

CONTACTS AND LOCATIONS:
Overall Officials: Helle Agger-Nielsen, dr., Principal Investigator — SVS - Sydvestjysk sygehus, Øre, næse og hals afdelingen
Locations (1):
- Hospital South West Jutland, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
Protocol review done by SDU (South Danish University)